CLINICAL TRIAL: NCT02038400
Title: Evaluation of the Efficiency of KINETUBE® in the Recurrent Chronic Tubal Ear Otitis Care (Otitis Media With Effusion, Atelectatic Otitis or Retraction) in Children With an Age Range of 7-15 Years.
Brief Title: Efficacy of KNT® (KINETUBE) in Recurrent Chronic Otitis Media in Children
Acronym: KINETUBE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-A00490-45; 2013-17 (Other: AP-HM)
Record Dates: First submitted 2013-11-28; First posted 2014-01-16 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2013-03

CONDITIONS: Chronic Otitis Infections in pédiatric Patients
MeSH Terms: interventions — Middle Ear Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group A (Experimental): KINETUBE medical Device
  Interventions: Device: insertion of tympanic ventilation tubes (tympanostomy)
- group B (Active Comparator): insertion of tympanic ventilation tubes (tympanostomy)
  Interventions: Device: KINETUBE medical Device

INTERVENTIONS:
Device: KINETUBE medical Device
  Arms: group B
Device: insertion of tympanic ventilation tubes (tympanostomy)
  Arms: group A

SUMMARY:
Otitis media are the consequence of bacterial infection. They are characterized by middle ear inflammations with a collection of fluid behind the eardrum. The effusion stagnates in the middle ear, can increase acute infection and induce tympanic membrane and inner ear damages. Delay in language learning can be observed in affected children as well as hearing problems e.g. constant hearing loss. The two main forms of chronic otitis are otitis media with effusion (OME) and atelectasis with or without retraction pockets.

To date, insertion of tympanic ventilation tubes (tympanostomy) is the most effective treatment for otitis media with effusion that has failed to respond to conservative drug treatments; and for delaying the progression of serious atelectasis. When a first tube did not allow complete recovery, recurrence is then observed and insertion of new tube is needed. The repeated tube insertions increase risks linked to general anesthesia and increase rate of sequelae/complications, such as tympanic membrane perforation.

Kinetube® is a CE-marked medical device, marketed in France and Europe since April 2002. This device improves the neuronal control mechanism of the pharyngotympanic (Eustachian) tube, regulating middle ear pressure. This could be an alternative for patients having recurrence and needing repeated tube insertion, as studies had shown that Kinetube® improved the opening of the Eustachian tube in patients with otitis media with effusion (OME) and atelectasis.

These previous clinical studies have shown the feasibility of the use of Kinetube® in clinical practice. A larger clinical study with a high level of evidence must be performed to show therapeutic efficacy of the Kinetube® in chronic otitis compared to ventilation tube insertion.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 7 to 15 years old
* Patients presenting recurrent otitis media with effusion, or atelectasis (with or without retraction pocket), with presence of fluid behind the eardrum, and conductive hearing loss ≥ 30 dB
* Patients who had undergone one (or more) previous tympanoplasty tube insertion, and who need a new one
* Patients whose parents (or parental authority holders) have given voluntary signed informed consent
* Patients affiliated to the French health insurance system or similar

Exclusion Criteria:

* Age less than 7 years old and higher than 15 years old
* Patients needing tympanoplasty tube insertion for the first time
* Patients who had already received Kinetube® treatment
* Patients presenting purulent acute otitis media
* Patients presenting otitis media with effusion following barotrauma
* Patients presenting neck dysfunction (cleft lip and cleft palate)
* Patients presenting nasopharynx and nasal cavities tumoral process (except adenoids)
* Patients with a narrow ear canal that does not allow tympanometry exam
* Patients with a history of irradiation of the ear, nose and throat
* Patient who underwent a previous surgery of the soft palate, or with paralysis of the soft palate
* Patients presenting cilia-related disease or chronic immunodeficiency
* Patients with Down syndrome
* Patients taking part, or having taken part, into other clinical study for the treatment of chronic otitis media

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2013-11; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Difference of the deficiency of hearing | 3 years
  Difference of the deficiency of hearing(audition) in decibels HL ( Hearing Level), measured by examination of tonal audiometry (average of the losses in air conductions with the frequencies 500-1000-2000 Hz), between the inclusion and 12 months after the implementation of the treatment(processing)

CONTACTS AND LOCATIONS:
Overall Officials: LOIC MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France